CLINICAL TRIAL: NCT01463735
Title: Vitamin E Supplement in Patients With Cirrhosis and Acanthocytosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Laurent Spahr, Principal Investigator, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CER 10-099
Record Dates: First submitted 2011-10-19; First posted 2011-11-02 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Cirrhosis
Keywords: Cirrhotic patients
MeSH Terms: conditions — Fibrosis | interventions — tocophersolan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Vitamin E supplement (tocofersolan) — 700 mg per day per os (i.e. 350 mg twice a day with meals)

SUMMARY:
Acanthocytes, also termed spur cell, are large erythrocytes covered with spike-like projections which are associated with severe hemolytic anemia. In advanced cirrhosis, acanthocytes may account for 20 to 30% of red blood cells. Up to 70% of cirrhotic patients display anemia and hemoglobin level may fall to below 5 gr/L in spur cell anemia. The true incidence of spur cells in cirrhosis is not known precisely but may avoisinate 45%, typically in patients with advanced cirrhosis.The presence of spur cells usually predicts lower survival rates. Vitamin E is an antioxidant compound that is a component of biological membrane that helps to maintain integrity of lipid bilayers. Vitamin E deficiency leads to erythrocyte hemolysis, which is improved by supplemental vitamin E. This study is an open label single arm phase II study in cirrhotic patients treated for 4 weeks with Tocofersolan (Vedrop), a water-soluble derivative of alpha-tocopherol, and thus an orally bio-available source of vitamin E. The aim of this study is to determine the effect of tocofersolan on red blood cell membranes lipid composition in adult patients with cirrhosis and vitamin E deficiency. Secondary endpoints are the effects of tocofersolan on anemia, hemolysis and acanthocytosis; on lipid peroxidation and oxidative stress; the safety of a 4 week treatment of 700 mg/day.

DETAILED DESCRIPTION:
Background:

Cirrhosis may be complicated by the presence of ascites, portosystemic collaterals that may eventually bleed or give rise to hepatic encephalopathy. Laboratory findings in patients with cirrhosis includes alterations in synthetic function as well as an increase in serum bilirubin. Liver diseases are also associated with hematologic complications and altered red blood cells morphology. Up to 70% of cirrhotic patients display anemia and hemoglobin level may fall to below 5 gr/L in spur cell anemia. Thrombocytopenia, leucopenia and neutropenia are also common. In patients with cirrhosis, acanthocytes and echinocytes are reported. Acanthocytes, also termed spur cell, are large erythrocytes covered with spike-like projections which are associated with severe hemolytic anemia. In advanced cirrhosis, acanthocytes may account for 20 to 30% of red blood cells. The spiky morphology of acanthocytes results from an abnormal surface area to volume ratio and an altered membrane lipids composition. These changes in red blood cell membranes render the cell more prone to destruction and hemolysis. The true incidence of spur cells in cirrhosis is not known precisely but may avoisinate 45%, typically in patients with advanced cirrhosis.The presence of spur cells usually predicts lower survival rates. The liver is a very susceptible organ to oxidative-related cellular damage, and low antioxidants, such as vitamin E, in cirrhosis participate in cellular membrane alterations. Vitamin E is an antioxidant compound that is a component of biological membrane that helps to maintain integrity of lipid bilayers. Vitamin E deficiency leads to erythrocyte hemolysis, which is improved by supplemental vitamin E. Tocofersolan (Vedrop) is a water-soluble derivative of alpha-tocopherol, and thus an orally bio-available source of vitamin E. Vitamin E supplementation appears safe in liver diseases and provides histological benefit in NASH.

Aim and endpoints I. To determine the effect of tocofersolan on red blood cell membranes lipid composition in adult patients with cirrhosis and vitamine E deficiency II. To determine the effect of vit E on anemia, hemolysis and acanthocytosis; on lipid peroxidation and oxidative stress; the safety of a 4 week treatment of 700 mg/day

Duration: selection period: 1 week; active treatment: 4 weeks; follow-up period. 3 weeks. Evaluation time-points: baseline and after 4 weeks of treatment Methodology/Design: phase II pilot trial on 27 patients, single arm study

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Cirrhosis (histology or, if not available, based on clinical, biological and radiological findings)
* Total bilirubin > 60 µmol/ L
* Anemia defined as hemoglobin < 120 g/L
* Vitamin E deficiency as defined by plasma levels < 23 µmol/L

Exclusion Criteria:

* Inability or unwillingness to give written consent
* Parenteral nutrition
* Co-medication with Orlistat, Colestipol, anticoagulants
* Active alcohol consumption as assessed by urine analysis
* Gastro-intestinal bleeding within the past 2 weeks
* Gastric bypass
* Moderate to severe renal failure as defined by creatinine clearance < 60 ml/min
* Hypothyroidism as defined by TSH > 6 mU/L
* Diagnosis of cancer upon inclusion in the study
* Any other severe condition affecting interfering with the normal conduct of the study
* Already participating in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
C/P (cholesterol to phospholipid) ratio of erythrocyte membrane before and after tocofersolan | 8 weeks

SECONDARY OUTCOMES:
percentage of acanthocytes in peripheral blood before and after tocofersolan | 8 weeks
plasma levels of vit E before and after tocofersolan | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals, Geneva, Switzerland